CLINICAL TRIAL: NCT00001322
Title: The Central Nervous System Effects of Pharmacologically Induced Hypogonadotropic Hypogonadism With and Without Estrogen and Progesterone Replacement
Brief Title: The Effects of Reproductive Hormones on Mood and Behavior
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: 920174; 92-M-0174
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2022-02-24 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2021-02-25

CONDITIONS: Healthy Volunteers
Keywords: Behavior; Brain Function; Progesterone; Central Nervous System Function; gonadotropin-releasing hormone (GnRH) Agonist
MeSH Terms: conditions — Behavior | interventions — Estradiol; Progesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 - Lupron (Experimental): Eight to 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly.
  Interventions: Drug: Leuprolide Acetate 3.75
- Phase 2, Arm 1 - Estradiol, then progesterone (Experimental): 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Additionally, 4 weeks of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 5 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day). Followed by 1-2 weeks (weeks 6-7) washout period. Then crossover to 5 weeks (week 8-12) of Progesterone suppositories (200mg vaginally twice/day) and placebo patches.
  Interventions: Drug: Leuprolide Acetate 3.75; Drug: Estradiol; Drug: Progesterone; Drug: Placebo suppository; Drug: Placebo patch
- Phase 2, Arm 2 - Progesterone, then estradiol (Experimental): 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly. Additionally, 5 weeks of Progesterone suppositories (200mg vaginally twice/day) and placebo patches. Followed by 1-2 weeks (weeks 6-7) washout period. Then crossover to 4 weeks (weeks 8-11) of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 12 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day).
  Interventions: Drug: Leuprolide Acetate 3.75; Drug: Estradiol; Drug: Progesterone; Drug: Placebo suppository; Drug: Placebo patch

INTERVENTIONS:
Drug: Leuprolide Acetate 3.75 — Eight to 12 weeks of GnRH agonist, Leuprolide Acetate 3.75 mg given intramuscularly monthly
Drug: Estradiol — Transdermal Estradiol, 100mcg/day by skin patch
  Arms: Phase 2, Arm 1 - Estradiol, then progesterone; Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Progesterone — Progesterone suppository, 200mg vaginally twice/day
  Arms: Phase 2, Arm 1 - Estradiol, then progesterone; Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Placebo suppository — Placebo suppository twice daily
  Arms: Phase 2, Arm 1 - Estradiol, then progesterone; Phase 2, Arm 2 - Progesterone, then estradiol
Drug: Placebo patch — Placebo by skin patch
  Arms: Phase 2, Arm 1 - Estradiol, then progesterone; Phase 2, Arm 2 - Progesterone, then estradiol

SUMMARY:
This study evaluates the effects of estrogen and progesterone on mood, the stress response, and brain function in healthy women.

The purpose of this study is to evaluate how low levels of estrogen and progesterone (that occur during treatment with leuprolide acetate) compare to menstrual cycle levels of estrogen and progesterone (given during individual months of hormone add-back) on a variety of physiologic measures (brain imaging, stress testing, etc.) in healthy volunteer women without PMS.

This study will investigate effects of reproductive hormones by temporarily stopping the menstrual cycle with leuprolide acetate and then giving, in sequence, the menstrual cycle hormones progesterone and estrogen. Tests (such as brain imaging or stress testing, etc.) will be performed during the different hormonal conditions (low estrogen and progesterone, progesterone add-back, estrogen add-back). The results of these studies will be compared between women without PMS and women with PMS (see also protocol 90-M-0088).

At study entry, participants will undergo a physical examination. Blood, urine, and pregnancy tests will be performed. Cognitive functioning and stress response will be evaluated during the study along with brain imaging and genetic studies.

DETAILED DESCRIPTION:
Evidence suggests that the gonadal steroids may exert clinically significant effects on central nervous system function. For example, the menstrual cycle may influence the occurrence of seizures in some female epileptics and the performance on certain cognitive tests. Central nervous system effects of gonadal steroids have been inferred largely from changes in behavior occurring in association with presumed changes in gonadal steroids during the normal menstrual cycle, during the administration of ovarian hormones, or in a gender-specific context. These inferences are, by definition, indirect and associational in nature and further are incapable of disentangling the effects of hormones which are simultaneously present in women of reproductive age. This study is designed to address those problems by comparing measures during Lupron-induced hypogonadism with those during replacement with estrogen or progesterone. On the basis of prior findings from our group and from others, we will be asking the following questions: 1) Is the decreased r-CBF that we observed in the prefrontal cortex during the hypogonadal state confirmed in individual women using new imaging techniques; 2) Will variation in genotype (e.g., COMT val/met, BDNF val/met) confer differential sensitivity to ovarian steroids in brain circuitry and 3) Are the menstrual cycle phase-related changes in reward systems that we previously observed related to estradiol or progesterone actions within the brain (1). Additionally, this protocol will serve as a control study for protocol # 90-M-0088.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers participating in this study will be women meeting the following criteria:

Between the ages of 18 and 50 years,

Not pregnant,

In good medical health,

Medication free,

No history of menstrual-related mood or behavioral disturbances.

Additionally, we will recruit a subsample of 20 asymptomatic women who will meet all inclusion and exclusion criteria in this protocol except they will have a history of a past major depressive episode.

Finally, a third sample of 10 women who meet all the inclusion and exclusion criteria listed above for this protocol will be recruited to establish the dose range of transdermal estrogen gel for this and related protocols (i.e., 90-M-0088 and 05-M-0059).

EXCLUSION CRITERIA:

The following conditions will constitute contraindications to treatment with hormonal therapy and will preclude a subject's participation in this protocol:

Current Axis I psychiatric diagnosis (with the exception of this women with a past major depression who will be studied on this protocol);

History consistent with endometriosis;

Diagnosis of ill-defined, obscure pelvic lesions, particularly undiagnosed ovarian enlargement;

Hepatic disease as manifested by abnormal liver function tests;

History of mammary carcinoma;

History of pulmonary embolism or phlebothrombosis;

Undiagnosed vaginal bleeding;

Porphyria;

Diabetes mellitus;

History of malignant melanoma;

Cholecystitis or pancreatitis;

Cardiovascular or renal disease;

Pregnancy;

Any woman meeting the Stages of Reproductive Aging Workshop Criteria (STRAW) for the perimenopause (129). Specifically, we will exclude any woman with an elevated plasma follicle stimulating hormone (FSH) level (greater than or equal to 14 IU/L) and with menstrual cycle variability of > 7 days different from their normal cycle length.

National Institute of Mental Health (NIMH) employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Subjects taking birth control pills will be excluded from the study.

Subjects taking diuretics, prostaglandin inhibitors, or pyridoxine (putative treatments for MRMD) will similarly be excluded from the study, as will patients taking psychotropic agents (e.g., lithium carbonate, tricyclic antidepressants).

All subjects will be required to use non-hormonal forms of birth control (e.g., barrier methods) to avoid pregnancy during this study.

Participants who have an active condition that places them at an increased risk for osteoporosis will be excluded from this protocol.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 1994-06-09 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Burgess LH, Handa RJ. Chronic estrogen-induced alterations in adrenocorticotropin and corticosterone secretion, and glucocorticoid receptor-mediated functions in female rats. Endocrinology. 1992 Sep;131(3):1261-9. doi: 10.1210/endo.131.3.1324155.
- [Background] Berman KF, Schmidt PJ, Rubinow DR, Danaceau MA, Van Horn JD, Esposito G, Ostrem JL, Weinberger DR. Modulation of cognition-specific cortical activity by gonadal steroids: a positron-emission tomography study in women. Proc Natl Acad Sci U S A. 1997 Aug 5;94(16):8836-41. doi: 10.1073/pnas.94.16.8836. PMID 9238064
- [Derived] Li HJ, Goff A, Rudzinskas SA, Jung Y, Dubey N, Hoffman J, Hipolito D, Mazzu M, Rubinow DR, Schmidt PJ, Goldman D. Altered estradiol-dependent cellular Ca2+ homeostasis and endoplasmic reticulum stress response in Premenstrual Dysphoric Disorder. Mol Psychiatry. 2021 Nov;26(11):6963-6974. doi: 10.1038/s41380-021-01144-8. Epub 2021 May 25. PMID 34035477
- [Derived] Di Florio A, Alexander D, Schmidt PJ, Rubinow DR. Progesterone and plasma metabolites in women with and in those without premenstrual dysphoric disorder. Depress Anxiety. 2018 Dec;35(12):1168-1177. doi: 10.1002/da.22827. Epub 2018 Sep 5. PMID 30184299
- [Derived] Nguyen TV, Reuter JM, Gaikwad NW, Rotroff DM, Kucera HR, Motsinger-Reif A, Smith CP, Nieman LK, Rubinow DR, Kaddurah-Daouk R, Schmidt PJ. The steroid metabolome in women with premenstrual dysphoric disorder during GnRH agonist-induced ovarian suppression: effects of estradiol and progesterone addback. Transl Psychiatry. 2017 Aug 8;7(8):e1193. doi: 10.1038/tp.2017.146. PMID 28786978
- [Derived] Wei SM, Baller EB, Kohn PD, Kippenhan JS, Kolachana B, Soldin SJ, Rubinow DR, Schmidt PJ, Berman KF. Brain-derived neurotrophic factor Val66Met genotype and ovarian steroids interactively modulate working memory-related hippocampal function in women: a multimodal neuroimaging study. Mol Psychiatry. 2018 Apr;23(4):1066-1075. doi: 10.1038/mp.2017.72. Epub 2017 Apr 18. PMID 28416813
- [Derived] Dubey N, Hoffman JF, Schuebel K, Yuan Q, Martinez PE, Nieman LK, Rubinow DR, Schmidt PJ, Goldman D. The ESC/E(Z) complex, an effector of response to ovarian steroids, manifests an intrinsic difference in cells from women with premenstrual dysphoric disorder. Mol Psychiatry. 2017 Aug;22(8):1172-1184. doi: 10.1038/mp.2016.229. Epub 2017 Jan 3. PMID 28044059
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1992-M-0174.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were screen failures, 4 withdrew prior to start of study and 92 started and completed phase 1 the study. 10 participants did not proceed to phase 2 (crossover arm) of the study.
Period: Phase 1 - Lupron Only
Arm/Group | Phase 1 - Lupron | Phase 2, Arm 1 - Estradiol, Then Progesterone | Phase 2, Arm 2 - Progesterone, Then Estradiol
Started | 92 | 0 | 0
Completed | 92 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2, Period 1 - Crossover Phase
Arm/Group | Phase 1 - Lupron | Phase 2, Arm 1 - Estradiol, Then Progesterone | Phase 2, Arm 2 - Progesterone, Then Estradiol
Started | 0 | 42 | 40
Completed | 0 | 42 | 40
Not Completed | 0 | 0 | 0
Period: Phase 2, Period 2 - Crossover Phase
Arm/Group | Phase 1 - Lupron | Phase 2, Arm 1 - Estradiol, Then Progesterone | Phase 2, Arm 2 - Progesterone, Then Estradiol
Started | 0 | 42 | 40
Completed | 0 | 42 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 - Lupron: Eight to 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly before randomization to estradiol or progesterone arm in the crossover phase of the study.
Arm/Group | Phase 1 - Lupron
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 92
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 55
  More than one race | 1
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Beck Depression Inventory Score
Description: The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures the severity of symptoms accompanying depression. Each item has a minimum score of 0 and a maximum score of 3, with higher numbers consistent with more severe symptoms. The score of each item is summed to amount the overall BDI score, with a minimum score of 0 and a maximum score of 63. Higher BDI scores are consistent with more severe depression. Score of 16 or greater is consistent with clinical depression.
  Each participant completed the BDI every 2 weeks during each of the study phases (i.e., GnRH agonist alone, estradiol and progesterone) throughout the 6-month study. Outcome measures reported consist of the average of two BDI scores from each phase of the study: the last 4 weeks of the GnRH agonist alone (phase 1), during the 4-week long estradiol phase (phase 2: weeks 2 and 4 of estradiol) and the 4-week long progesterone phase (phase 2: weeks 2 and 4 of progesterone).
Time Frame: Phase 1: Weeks 6 and 8 or 10 and 12; Phase 2: Weeks 2 and 4 of estradiol or progesterone
Population: Analyses included comparison of mean BDI scores during each phase of the study
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Phase 2 - Estradiol: 4 weeks of transdermal Estradiol (100mcg/day by skin patch) and placebo suppositories. Week 5 involves 100mcg/day transdermal Estradiol and active Progesterone suppositories (200mg vaginally twice/day).
- Phase 2 - Progesterone: 5 weeks of Progesterone suppositories (200mg vaginally twice/day) and placebo patches.
Arm/Group | Phase 1 - Lupron | Phase 2 - Estradiol | Phase 2 - Progesterone
Number analyzed (Participants) | 92 | 82 | 82
Units on a scale | 1.4 (2.1) | 1 (2) | 1.1 (1.8)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Lupron: Eight to 12 weeks of GnRH agonist treatment 3.75 mg given intramuscularly monthly.
- Phase 2 - Estradiol: 4 weeks of transdermal Estradiol (100mcg/day by skin patch)
- Phase 2 - Progesterone: 5 weeks of Progesterone suppositories (200mg vaginally twice/day)
Arm/Group | Lupron | Phase 2 - Estradiol | Phase 2 - Progesterone
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 1/92 | 1/82 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lupron (N=92) | Phase 2 - Estradiol (N=82) | Phase 2 - Progesterone (N=82)
Breast fibroma (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lupron (N=92) | Phase 2 - Estradiol (N=82) | Phase 2 - Progesterone (N=82)
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT00001322/Prot_SAP_000.pdf